CLINICAL TRIAL: NCT05027542
Title: Comparison of Distally Based Sural Artery and Supramalleolar Flap for Coverage of Dorsum of Foot and Ankle Defects; A CROSS-SECTIONAL STUDY OF 53 PATIENTS
Brief Title: Comparison of Distally Based Sural Artery and Supramalleolar Flap for Coverage of Dorsum of Foot and Ankle Defects
Status: Completed | Type: Observational
Sponsor: Abeer Musaddiq (Other)
Responsible Party: Sponsor-Investigator, Abeer Musaddiq, Research Officer, Aga Khan University Hospital, Pakistan
Organization: Aga Khan University Hospital, Pakistan (Other)
Other Study IDs: 4452
Record Dates: First submitted 2021-08-23; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Open Wound of Lower Limb
Keywords: Soft Tissue Injuries, fasciocutaneous flaps, Survival Rate
MeSH Terms: conditions — Soft Tissue Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our main aim for this study was to evaluate the long-term outcome comparisons between sural artery and Supramalleolar flap in the reconstruction of extensive defects of non-weight bearing regions of foot and ankle. The patients' information were collected through medical records and analyzed through SPSS

DETAILED DESCRIPTION:
In this article we intend to present our experience comparing a series of the two types of flaps in terms of viability, coverage of defect, cosmetic appearance, and functions of foot and ankle based on self-designed Tool . This Tool contains 4 parameters i.e., Activity of daily living, coverage of defect, cosmetic appearance of Skin post flap, and Weight bearing status. A score was given to each parameter and on the basis of these scores, Long term outcome were analyzed of each patient

ELIGIBILITY:
Inclusion Criteria:

* Only defects of foot and ankle around dorsum and perimalleolar areas were included.

Exclusion Criteria:

* The defects reconstructed with other local flaps and free flaps were excluded from this review

Ages: 2 Months to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data of all those patients was collected who underwent reconstruction of soft tissue defects of foot and ankle with Supramalleolar and sural artery flaps between 1996 and 2020. The data of these patients were collected from the Hospital inpatient management system and review of medical records through a structured proforma that included demographic variables, cause of soft tissue defects (secondary to open fractures, following debridement of chronic infected wounds, tumor excision and defects following release of scar contractures), side of defects, size and type of flap (supramalleolar or sural artery), complications and long-term outcome of the flap.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
self-designed assessment tool | 1996-2020
  The functional outcome of each patient was measured by activity of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Pervaiz Hashmi, Principal Investigator — Agha Khan University Hospital
Locations (1):
- Agha Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
data of study participants is only accessible to researcher of this study

DOCUMENTS (1):
  • Informed Consent Form (2020-11-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT05027542/ICF_000.pdf